CLINICAL TRIAL: NCT05386628
Title: The Effect of Myofascial Chain Release Techniques on Shoulder Joint Range of Motion Following Mastectomy Surgery in Breast Cancer Survivors
Brief Title: The Effect of Myofascial Chain Release Techniques on Shoulder Joint Range of Motion in Breast Cancer Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Nilufer Kablan, Head of Department, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022/0132
Record Dates: First submitted 2022-05-18; First posted 2022-05-23 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Breast Cancer Survivors
Keywords: breast cancer; range of motion; lymphatic drainage
MeSH Terms: conditions — Breast Neoplasms | interventions — Manual Lymphatic Drainage

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- control group (Active Comparator): Conventional physiotherapy program (joint movement exercises, local relaxation techniques, etc.) will be applied to the participants in this group.
  Interventions: Other: conventional physiotherapy
- Manual lymphatic drainage group (Experimental): In addition to the conventional physiotherapy program, manual lymphatic drainage (including upper limb extremity and anterior/posterior axillar-axillar anastomoses and axilla-inguinal anastomosis) will be applied to the participants in this group.
  Interventions: Other: conventional physiotherapy; Other: Manual lymphatic drainage
- Myofascial relasing group (Experimental): In addition to the conventional physiotherapy program, myofascial chain relasing techniques will be applied to the participants in this group.
  Interventions: Other: conventional physiotherapy; Other: Myofascial relasing
- Lymphatic drainage and myofascial releasing group (Experimental): In addition to the conventional physiotherapy program, manual lymphatic drainage (including upper limb extremity and anterior/posterior axillar-axillar anastomoses and axilla-inguinal anastomosis) and myofascial chain relasing techniques will be applied to the participants in this group.
  Interventions: Other: conventional physiotherapy; Other: Manual lymphatic drainage; Other: Myofascial relasing

INTERVENTIONS:
Other: conventional physiotherapy — A basic physiotherapy program consisting of shoulder exercises will be applied to the participants.
  content of the physiotherapy program
  * Shoulder passive/active abduction, flexion, internal and external rotation exercises
  * Posture exercises
  * Neck stretching exercises
  * Pectoralis major stretching exercises
  * Shoulder capsule stretching exercises
  * Scapular Mobilization exercises
Other: Manual lymphatic drainage — manual lymph drainage is a manual technique that is applied to the lymphatic system with a pressure of 40-50 mmHg and increases the working speed of lymphatic nodules/collectors. Manual lymph drainage will be made to the anterior axillar-axillar, posterior axillar-axillar and axilla-inguinal anastomosis collectors and the arm region (up to the elbow) lymph collectors.
  Arms: Lymphatic drainage and myofascial releasing group; Manual lymphatic drainage group
Other: Myofascial relasing — it will be done with the thumb or 3rd finger from the acu points of the superficial arm-anterior myofascial chain. 6-8 seconds with thumb to these points. pressure will be applied and vibration will be given clockwise.
  Arms: Lymphatic drainage and myofascial releasing group; Myofascial relasing group

SUMMARY:
In breast cancer patients, limitation of shoulder joint movement occurs following mastectomy surgery. Studies have reported that damage to the fascia on the pectoralis major muscle during mastectomy surgery contributes to the development of the limitation. The aim of this study is to investigate the effect of release techniques applied to the fascia on the pectoralis major muscle and the fascial chain on the incerasing of shoulder joint range of motion.

DETAILED DESCRIPTION:
After mastectomy, complications such as decreased range of motion and muscle strength in the shoulder joint, development of pain and tenderness, and formation of lymphedema are frequently observed. In addition to causing a significant decrease in the patient's daily life quality, shoulder limitation also negatively affects the treatment process by preventing the joint position required for radiotherapy. For this reason, it is a priority to prevent the development of shoulder joint limitations that may occur following surgery and to open the developing limitation immediately. This study was born from the idea that the relaxation techniques to be applied to regain the mobility of the fascial structure, which has been damaged and whose mobility has decreased due to breast surgery, should be performed by covering the entire myofascial chain. In addition, the investigators aim to prevent adhesions that will limit the mobility of soft tissue by minimizing scar tissue formation with early drainage of postoperative edema. The aim of this study is to investigate the effectiveness of myofascial chain relaxation techniques and manual lymphatic drainage applied to improve soft tissue mobility in the prevention and elimination of shoulder limitations after breast cancer surgery.

A total of 48 patients who agreed to participate in the study will be enrolled in the treatment program twice a week for 6 weeks. During the study, the same assessments will be applied to all patients and the cases will be evaluated 3 times (pre-treatment, post treatment, and one month post treatment). During the assessments, the physical evaluations of the patients on the shoulder region will be examined in detail using objective and subjective methods.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 30-60
* Having breast surgery within 2 years
* Not have received conservative treatment for shoulder rehabilitation in the last 6 months
* Having limitation of movement of the shoulder joint due to breast surgery

Exclusion Criteria:

* Not having agreed to participate in the study
* Having undergone radical mastectomy surgery
* Having connective tissue disease
* Presence of brachial plexus paresis/plegia
* Presence of radiogenic fibrosis
* Presence of additional orthopedic (scoliosis, etc.), neurological (multiple sclerosis, stroke, etc.) and rheumatological diseases (ankylosing spondylitis, rheumatoid arthritis, etc.) that will affect upper extremity functions
* Presence of active metastases
* Having undergone reconstruction surgery
* Continuation of radiotherapy (must have ended at least 3 months ago) or chemotherapy applications
* Having had a bilateral mastectomy
* To develop lymphedema in the arm-trunk
* Use of muscle relaxants
* Patients with severe chemotherapy side effects (hyperesthesia, nausea, skin changes, weakness, etc.)

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — breast cancer survivors
Enrollment: 48 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
measurement of tissue stiffness (N/m) | changes from baseline stiffness values will be measured at 6 week and 10 week
  Stiffness values will be measured with myotonPro on centers of coordination located along the myofascial chain .
measurement of passive muscle tone (Hz) | changes from baseline tone values will be measured at 6 week and 10 week
  muscle tones will be measured with myotonPro on centers of coordination located along the myofascial chain
measurement of creep of tissue | changes from baseline creep values will be measured at 6 week and 10 week
  creep of tissue will be measured with myotonPro on centers of coordination located along the myofascial chain
measurement of the range of shoulder joint motion | changes from baseline range of the shoulder joint motion values will be measured at 6 week and 10 week
  The range of shoulder flexion, abduction, extension and external-internal rotation movements will be measured with a universal goniometer.
assessment of activity of daily living | changes from baseline Quick-DASH Questionnaire scores will be assessment at 6 week and 10 week
  upper extremity daily living functional capacity of participation will be assessed with the Quick-DASH (Shortened Disabilities Arm, Shoulder and Hand Questionnaire). The scale consists of 11 items. In the scale, a 5-point Likert scale is evaluated and scored 1-5. The scores that can be obtained from the scale are between 0-100. Lower scores indicate better daily activity participation.
assessment of depression and anxiety | changes from baseline HAD scale scores will be assessment at 6 week and 10 week
  quality of life will be assessed using the Hospital Anxiety and Depression Scale (HAD). The scale consists of 14 items (7 items depression and 7 items anxiety). The scale is evaluated on a 4-point Likert scale and is scored 0-3. Depression and anxiety scores are calculated separately. While the score range that can be taken in the lower scales is 0-21, low scores are considered positive.

SECONDARY OUTCOMES:
measurement of skin temperature | changes from baseline skin temperature values will be measured at 6 week and 10 week
  measurements will be taken from the area covering 3 cm of the surgical incision with a P45 thermographic camera with high thermal sensitivity (Flir Sistem, ThermaCAM, Sweden).
measurement of pain | changes from baseline pain values will be measured at 6 week and 10 week
  Pain will be evaluated by visual analog scale (VAS). In the scale, the patient is asked to mark the most appropriate pain intensity on a scale ranging from 0 (no pain) to 10 (tolerable pain). The higher the score, the greater the pain intensity.
measurement of pain pressure threshold | changes from baseline pain pressure threshold values will be measured at 6 week and 10 week
  Pain pressure threshold will be evaluated by a digital algometer (Algometer Commander, Jtech Medical, MM036_K, 2016).
measurement of grip strength | changes from baseline grip strength values will be measured at 6 week and 10 week
  The grip strength of both hand will be evaluated by "hand-held" dynamometer.

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul Medeniyet University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: Individual Participant Data Set: 26079868 — https://pubmed.ncbi.nlm.nih.gov/
- Available data/document: Individual Participant Data Set: 16225693 — https://pubmed.ncbi.nlm.nih.gov/
- Available data/document: Individual Participant Data Set: 12924842 — http://pubmed.ncbi.nlm.nih.gov/
- Available data/document: Individual Participant Data Set: 31864435 — http://pubmed.ncbi.nlm.nih.gov/
- Available data/document: Individual Participant Data Set: 22018755 — http://pubmed.ncbi.nlm.nih.gov/
- Available data/document: Individual Participant Data Set: 18192154 — http://pubmed.ncbi.nlm.nih.gov/
- Available data/document: Individual Participant Data Set: 25977305 — http://pubmed.ncbi.nlm.nih.gov/
- Available data/document: Individual Participant Data Set: 20068255 — http://pubmed.ncbi.nlm.nih.gov/